CLINICAL TRIAL: NCT06997237
Title: The Effect of Music Played to Liver Transplant Donors During Surgery on Hemodynamic Parameters and Cortisol Levels: A Randomized Controlled Trial
Brief Title: The Effect of Music Played to Liver Transplant Donors During Surgery on Some Hemodynamic Values and Cortisol Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan SARITAŞ (Other)
Responsible Party: Sponsor-Investigator, Hasan SARITAŞ, Assistant Professor, Siirt University
Organization: Siirt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SARITAS-MUSIC01
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Surgical Stress Response
Keywords: Music Therapy; Cortisol; Hemodynamic Parameters; Liver Transplantation; Intraoperative Stress

STUDY DESIGN:
Intervention Model Description: This study employed a parallel assignment interventional model. Participants were randomly divided into three groups: (1) the music group, which received classical music intervention during surgery, (2) the silence group, which used noise-canceling headphones without music, and (3) the control group, which received no intervention. All participants were liver transplant donors. The hemodynamic values and cortisol levels of participants were measured and compared before, during, and after surgery to evaluate the physiological effects of music exposure.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Group (Experimental): Participants in this group listened to a playlist composed of music pieces they selected prior to surgery, consisting of approximately 5-6 tracks. The music was played continuously for 30 minutes during the surgery through Bluetooth headphones. The sound level was set at 65 decibels.
  Interventions: Behavioral: Music Listening Intervention
- Silence Group (Sham Comparator): Participants in this group wore headphones during the surgery, but no music was played. The headphones were used to block ambient operating room sounds. This group was used to control for the effect of wearing headphones without auditory stimulation.
  Interventions: Behavioral: Silence with Headphones
- Control Group (No Intervention): Participants in this group did not receive any intervention. No headphones were worn, and no music or auditory stimulus was provided during the surgery. This group served as the control to compare the effects of music and silence interventions.

INTERVENTIONS:
Behavioral: Music Listening Intervention — Participants listened to a playlist of 5-6 music tracks they personally selected before surgery. The music was played continuously for 30 minutes through Bluetooth headphones during liver transplantation. Volume was kept at 65 decibels.
  Arms: Music Group
Behavioral: Silence with Headphones — Participants wore Bluetooth headphones during the surgery, but no audio was played. This intervention was designed to control for the effect of wearing headphones and isolating ambient operating room sounds.
  Arms: Silence Group

SUMMARY:
This randomized controlled trial investigates the effects of music played during liver donor surgery on hemodynamic parameters and cortisol levels. Ninety participants were divided into three groups: music, silence (with headphones but no sound), and a control group with no intervention. The study aimed to evaluate whether music can reduce stress-related physiological responses during surgery.

DETAILED DESCRIPTION:
This study was designed to evaluate the effects of music played during surgery on liver transplant donors. The research included 90 adult participants who underwent live liver donation surgeries. Participants were randomly assigned to one of three groups: music group (headphones with music), silence group (headphones without sound), and a control group (no headphones). Music intervention lasted for 30 minutes during the operation.

The primary objective was to examine whether intraoperative music exposure could reduce physiological stress, measured via cortisol levels. Secondary outcomes included changes in hemodynamic parameters such as systolic and diastolic blood pressure, pulse rate, oxygen saturation, and respiratory rate. Measurements were taken before and after the surgery.

The study was conducted at İnönü University Liver Transplant Institute, with ethical approval granted by the Malatya Clinical Research Ethics Committee (Approval No: 2021/52). The findings suggest that music may be an effective supportive intervention for reducing surgical stress.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years

Undergoing elective surgery as a liver donor

No physical or mental condition preventing listening to music

Willing to participate voluntarily and signing the informed consent form

Exclusion Criteria:

* Development of hemodynamic instability during anesthesia induction

Participants for whom the study could not be continued due to technical reasons during surgery

Participants who did not comply with the study protocol or had incomplete records

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Serum Cortisol Levels During the Intraoperative Period | Intraoperative (from pre-induction to the 30th minute of surgery)
  Serum cortisol levels were measured at two intraoperative time points: (1) immediately before anesthesia induction and (2) at the 30th minute of surgery. Blood samples were drawn from the radial artery, centrifuged, stored at -80°C, and later analyzed using the ELISA method. The difference between the two measurements was calculated to evaluate the physiological impact of the interventions.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure During the Intraoperative Period | Intraoperative (from pre-induction to the 30th minute of surgery)
  Systolic blood pressure was measured at two intraoperative time points: (1) immediately before anesthesia induction and (2) at the 30th minute of surgery. The difference between the two values was used to assess the hemodynamic effect of music and silence interventions compared to standard care.
Change in Diastolic Blood Pressure During the Intraoperative Period | Intraoperative (from pre-induction to the 30th minute of surgery)
  Diastolic blood pressure was measured at two intraoperative time points: (1) immediately before anesthesia induction and (2) at the 30th minute of surgery. Blood pressure was monitored continuously using a non-invasive automated device. The difference between the two values was analyzed to assess the effects of music and silence interventions on intraoperative hemodynamic response.
Change in Heart Rate During the Intraoperative Period | Intraoperative (from pre-induction to the 30th minute of surgery),
  Heart rate was recorded at two intraoperative time points: (1) immediately before anesthesia induction and (2) at the 30th minute of surgery. Monitoring was performed using standard intraoperative ECG. The difference between the two values was analyzed to evaluate the effect of music and silence interventions on autonomic cardiac response during surgery.
Change in Respiratory Rate During the Intraoperative Period | Intraoperative (from pre-induction to the 30th minute of surgery)
  Respiratory rate was recorded at two intraoperative time points: (1) immediately before anesthesia induction and (2) at the 30th minute of surgery. Monitoring was conducted using standard intraoperative vital sign monitoring systems. The difference between the two values was analyzed to evaluate the effect of music and silence interventions on respiratory function.
Change in Peripheral Oxygen Saturation (SpO₂) During the Intraoperative Period | Intraoperative (from pre-induction to the 30th minute of surgery)
  Peripheral oxygen saturation (SpO₂) was measured at two intraoperative time points: (1) immediately before anesthesia induction and (2) at the 30th minute of surgery. Measurements were taken using standard pulse oximetry. The difference between the two values was used to assess the impact of music and silence interventions on tissue oxygenation during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Meral ÖZKAN, Prof. Dr., Study Chair — Inonu University Faculty of Nursing
Locations (1):
- Turgut Özal Medical Center, Liver Transplantation Institute, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study did not include a plan for data sharing in the ethical approval and informed consent process. Participant confidentiality and data protection are prioritized.